CLINICAL TRIAL: NCT05690204
Title: A Phase 2B Double-blind, Placebo-controlled, Dose-finding Study to Evaluate the Efficacy and Safety of 3 Dosages of SAP-001 in Combination With Standard of Care in Adult Subjects With Gout
Brief Title: Dose Finding Study to Evaluate Safety and Efficacy of 3 Dosages of SAP 001.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanton Pharma Pte. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAP-001-202
Record Dates: First submitted 2022-12-12; First posted 2023-01-19 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Gout
Keywords: Hyperuricemia; Serum Uric Acid; Gout Flare
MeSH Terms: conditions — Gout; Hyperuricemia | interventions — Colchicine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo versus SAP-001 (Experimental): Placebo arm
  Interventions: Drug: SAP-001
- SAP-001 low dose (Experimental): SAP-001 low dose
  Interventions: Drug: SAP-001
- SAP-001 middle dose (Experimental): SAP-001 middle dose
  Interventions: Drug: SAP-001
- SAP-001 high dose (Experimental): SAP-001 high dose
  Interventions: Drug: SAP-001

INTERVENTIONS:
Drug: SAP-001 — Test the efficacy and safety of SAP-001 versus placebo
  Other Names: Xanthine Oxidase Inhibitor; Colchicine

SUMMARY:
The aim of this study is to confirm the safety and pharmacological characteristics of SAP-001, evaluate its efficacy in lowering sUA and tophus burden, and identify the appropriate dose regimen for future studies in adult subjects with gout, with or without tophi, and hyperuricemia refractory to SoC XOI therapy.

DETAILED DESCRIPTION:
A Phase 2B, multicenter, randomized, double-blind, placebo-controlled, dose-finding study to assess the safety, PK, PD, and efficacy of 3 orally administered dosages of SAP-001 compared to placebo QD in adult subjects with gout, with or without tophi, and hyperuricemia refractory to standard-of-care (SoC) XOI therapy. In the completed Phase 1 and Phase 2 studies, SAP-001 was well tolerated at single doses up to 120 mg and at dosages up to 60 mg QD for 28-days in subjects with gout and hyperuricemia and demonstrated statistically significant reductions in sUA levels compared to placebo.

The aim of this study is to confirm the safety and pharmacological characteristics of SAP-001.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female, ≥18 and ≤75 years of age, willing and able to provide informed consent and to adhere to the requirements and guidelines of the protocol.
2. Body mass index ≥19 and ≤40 kg/m2 at the Screening Visit (Visit 1).
3. Already have been diagnosed with gout according to the current American College of Rheumatology (ACR) scoring criteria for the classification of primary gout; or has symptoms of gout with at least 1 of the following: i. 3 gout flares in the previous 18 months prior to screening; or ii. Presence of at least 1 gout tophus; or iii. Current diagnosis of gouty arthritis; Subject must be refractory to SoC XOI therapy, or in whom XOI is contraindicated. Refractory to SOC XOI is defined by a medical history of failure to normalize sUA to <6 mg/dL (the ACR target for gout) with at least 3 months of SoC XOI treatment at the maximum medically appropriate dose. XOI contraindication can be self-reported medical contraindication to SoC XOI therapy or in whom SoC XOI therapy is not considered medically appropriate treatment for symptomatic gout. Subject can still participate in the clinical trial if SOC XOI therapy is considered medically not appropriate or contraindicated.
4. Subject must have been on SoC XOI therapy for gout and hyperuricemia for at least 4 weeks immediately before the Randomization Visit (Day 1, Visit 4) unless SoC XOI therapy is contraindicated or not medically appropriate. Subjects who stopped SoC XOI therapy within 4 weeks of the Screening Visit are eligible for the study but must be restarted on SoC XOI therapy and confirmed resistant to XOI therapy (sUA levels ≥7.0 mg/dL) after at least 4 weeks of treatment.
5. Subject must have sUA levels ≥7.0 mg/dL by central laboratory results at the Screening Visit (Visit 1) and prior to randomization at the Randomization Visit (Day 1, Visit 4).

Main Exclusion Criteria:

1. Subjects not previously diagnosed as having gout before the Screening Visit.
2. Female subject is pregnant, planning to get pregnant, lactating/breastfeeding, or has a positive urine pregnancy test at the Screening Visit or prior to randomization at the Randomization Visit (Day 1, Visit 4).
3. Subject has used any prescription drugs (eg, losartan, pegloticase, URAT1 inhibitors), OTC medications, herbal medications or products, vitamins, or minerals that are known to lower sUA levels (except SoC XOI therapies) within 14 days prior to the Randomization Visit (Day 1, Visit 4). Exceptions may be made on a case-by-case basis (such as chronic use of low dose aspirin) following discussion and agreement between the investigator and sponsor. Subjects who are already taking losartan for blood-pressure control are allowed to enroll in the study and continue taking losartan if they have been on a stable dose for at least 6 months.
4. Subject was not compliant with taking placebo during the Run-in Period (defined as taking <80% or >120% of planned placebo doses) or the investigator determines that the subject was not compliant with SoC XOI gout medications (unless SoC XOI therapy is contraindicated or not medically appropriate) during the Run-in Period as assessed prior to randomization at the Randomization Visit (Day 1, Visit 4).
5. Subject had an acute gout flare (exclusive of symptomology associated with chronic synovitis/arthritis) that did not resolve at least 14 days prior to the Randomization Visit (Day 1, Visit 4). If an acute gout flare occurs during the Screening or Run-in Periods, the subject may be rescreened after a period of at least 14 days has passed following resolution of the flare.
6. Serum creatinine level >1.5 mg/dL and/or eGFR ≤60 mL/min/1.73 m2 calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation23 by central laboratory results at the Screening Visit (Visit 1) or prior to randomization at the Randomization Visit (Day 1, Visit 4).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
primary | 24 weeks
  assess the proportion of subjects who achieved sUA levels less than 6 mg/dl by laboratory results

SECONDARY OUTCOMES:
AE | 24 weeks
  Incidence of AEs including SAE and TEAEs by CTCAE criteria
Change from Baseline on PE measure | 24 weeks
  Changes from baseline in Physical Exam based on number of participants with abnormal findings
Changes from Baseline on ECGs | 24 weeks
  Changes from baseline in ECG parameters by QTc intervals

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Arencibia, Study Director — Study Official
Locations (15):
- United States (14):
  - California Site, Sacramento, California
  - California Site, San Diego, California
  - Denver Site, Denver, Colorado
  - Florida Site, DeBary, Florida
  - Florida Site, Miami, Florida
  - Florida Site, Miami Lakes, Florida
  - Florida Site, Winter Park, Florida
  - Idaho Site, Boise, Idaho
  - Maryland Site, Oxon Hill, Maryland
  - Mississippi Site, Jackson, Mississippi
  - North Carolina Site, Raleigh, North Carolina
  - Texas Site, Mesquite, Texas
  - Texas Site, Plano, Texas
  - Texas Site, The Woodlands, Texas
- Puerto Rico Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No